CLINICAL TRIAL: NCT06298994
Title: Kronik Obstrüktif Akciğer Hastalığında Vücut Farkındalığı, Fonksiyonel Hareket Analizi ve İlişkili Parametrelerin Belirlenmesi
Brief Title: Determination of Body Awareness and the Functional Movement in Patients With COPD
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, Principal investigator; PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: SBA 23/391
Record Dates: First submitted 2024-02-27; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Postural; Defect; Movement, Abnormal; Pain
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyskinesias; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: Patients with Chronic Obstructive Pulmonary Disease
- control group: Aged-matched healthy controls

SUMMARY:
The aim of this study is to investigate body awareness and functional movement in patients with Chronic Obstructive Pulmonary Disease (COPD) compared to healthy controls.

DETAILED DESCRIPTION:
It is aimed at investigating body awareness, and functional movement, and related factors in patients with COPD. The secondary purpose is to determine correlations between body awareness and functional movement, respiratory muscle strength and endurance, daily living activities, posture, and pain threshold in this study. The determination of correlations between functional movement, respiratory pattern, and functional exercise capacity is also purposed. In accordance with these purposes, at least 30 patients with COPD will be included and at least 30 healthy controls will be included. Tests and questionnaires will be used in order to determine the severity of disease. Lung function test and respiratory muscle strength and endurance test will be performed. Six Minute Walk Test will be performed for functional exercise capacity. To evaluate posture, the Corbin Postural Assessment Scale will be used. Pain and pain threshold will be assessed via Visual Analog Scale and an algometer, respectively. Body Awareness Rating Questionnaire will be used for evaluating body awareness. To evaluate daily living activities, Glittre Activities of Daily Living Test will be used. The Functional Movement Screen Test will be used for functional movement analysis. According to the results to be obtained, body awareness and functional movement will be determined in patients with COPD. It will guide professional working in this field.

ELIGIBILITY:
Inclusion Criteria for Chronic Obstructive Pulmonary Disease Group

* Being under 55 years old
* To be literate,
* Having volunteered to participate in the research,
* Stage 1-2-3-4 according to the Classification of Airflow Limitation in COPD (GOLD) system,
* Being clinically stable for the last 2 weeks.

Exclusion Criteria for Chronic Obstructive Pulmonary Disease Group

* Having history of lung cancer, sarcoidosis, tuberculosis and/or lung surgery,
* Communication problems,
* Having a severe psychiatric disorder.

Inclusion Criteria for Healthy Control Group

* Not having any cardiopulmonary system disease or chronic systemic disease,
* To be literate,
* Being under 55 years old
* Be willing to participate in the study.
* Not having balance problems, musculoskeletal, neurological and psychiatric disorders that could prevent performing the test procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with COPD and aged matched healthy controls will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-08 (Estimated); Primary Completion 2025-03-08 (Estimated); Study Completion 2026-03-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of functional movement | 1 day
  Functional movement analysis will be performed via The Functional Movement Screen.
Evaluation of Body Awareness | 1 day
  Body awareness will be assessed via Body Awareness Rating Questionnaire. It consists of 24 questions and each item is scored on a 7-point Likert-type scale. The total score ranges from 24 to168. A Higher scores indicate higher body awareness.

SECONDARY OUTCOMES:
Functional exercise capacity | 1 day
  Functional exercise capacity will be assessed via Six minute walk test.
Respiratory muscle strength | 1
  Respiratory muscle strength will be assessed via a using a mouth pressure device according to American Thoracic Society/ European Respiratory Society guidelines.
Respiratory muscle endurance | 1 day
  Respiratory muscle endurance will be assessed using the maximal incremental loading technique and constant loading technique using a device according to the European Respiratory Society guidelines.
Pain Severity | 1 day
  Severity of pain will be assessed via Visual Analog Scale. Zero point is defined as no pain and ten point as unbearable pain. Total point ranges from 0 to 10.
Pain threshold | 1 day
  Pain threshold will be assessed via an algometer.
Posture | 1 day
  Posture will be examined via the Corbin Postural Assessment Scale. The total points of the Corbin Postural Assessment Scale range from 0 to 28 points. A higher point represents worse posture.
Daily living activities | 1 day
  Daily living activities will be evaluated via Glittre Activities of Daily Living Test.
Severity of disease | 1 day
  Global Initiative for Chronic Obstructive Pulmonary Disease and Global Initiative for Chronic Obstructive Pulmonary ABE assessment Tool will be used for severity of disease. According to the Global Initiative for Chronic Obstructive Pulmonary Disease, the severity of airflow limitation (Forced Expiratory Volume in 1 s) was determined as mild (≥ 80%), moderate (50-80%), severe (30-50%), and very severe (<30%). According to Global Initiative for Chronic Obstructive Pulmonary A,B,E assessment Tool, patients classified group A, B, and E using symptom status and airflow limitation.
Dyspnea | 1 day
  The Modified Medical Research Council will be used for patients with COPD. The Modified Medical Research Council consist of five grades. A higher grades represents severe dyspnea level.
Symptoms | 1 day
  Chronic Obstructive Pulmonary Disease Assessment Test will be used to determine symptoms. The total score of Chronic Obstructive Pulmonary Disease Assessment Test changes from 0 to 40 points, and 10 points is the accepted cut-off point for COPD.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Aynur Demirel, Ankara
  - Hacettepe University, Ankara